CLINICAL TRIAL: NCT06152341
Title: Safety and Effectiveness of the ATC System in the Treatment of Acute Pulmonary Embolism
Brief Title: Safety and Effectiveness of the ATC System in the Treatment of Acute PE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akura Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-60003
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients with Acute Pulmonary Embolism (Experimental): Patients undergoing mechanical thrombectomy for acute pulmonary embolism.
  Interventions: Device: ATC System

INTERVENTIONS:
Device: ATC System — The ATC System is designed to mechanically remove emboli and restore blood flow through the pulmonary arteries in patients experiencing acute PE

SUMMARY:
This study is a prospective, single-arm, interventional, multicenter study to evaluate the safety and effectiveness of the ATC System in subjects with acute pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 and ≤ 90 years old
2. Clinical signs and symptoms consistent with acute PE for < 14 days
3. CTA evidence of proximal PE
4. RV/LV ratio > 0.9
5. Systolic BP ≥90 mmHg without the need for vasopressors
6. Stable heart rate (HR) < 130 BPM prior to procedure
7. Patient is deemed medically eligible for interventional procedure(s), per investigator guidelines and clinical judgment
8. Subject or legally authorized representative (LAR) is willing and able to provide written informed consent prior to receiving any non-standard of care protocol specific procedures

Exclusion Criteria:

1. Prior PE < 180 days from index procedure
2. Thrombolytic use < 30 days prior to baseline CTA
3. Pulmonary hypertension with peak pulmonary artery systolic pressure (PASP) >70 mmHg by right heart catheterization
4. FiO2 requirement >40% or >6 LPM to keep oxygen saturation >90%
5. Hematocrit <28%
6. Platelets count <100,000/µL
7. Serum creatinine >1.8 mg/dL
8. International normalized ratio (INR) >3
9. Major trauma injury severity score (ISS) >15 prior to screening assessment
10. Presence of intracardiac lead in right ventricle or atrium placed within 6 months prior to screening assessment
11. Cardiovascular or pulmonary surgery within 7 days of index procedure
12. Actively progressing cancer treated by chemotherapeutics
13. Known bleeding diathesis or coagulation disorder
14. Left bundle branch block
15. History of severe or chronic pulmonary arterial hypertension
16. History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
17. History of decompensated heart failure
18. History of underlying lung disease that is oxygen dependent
19. History of chest irradiation
20. History of heparin-induced thrombocytopenia (HIT)
21. Contraindication to systemic or therapeutic doses of anticoagulants
22. Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
23. Imaging evidence or other evidence that suggest, in the opinion of the investigator, the Subject is not appropriate for aspiration thrombectomy intervention
24. Life expectancy <90 days, as determined by investigator such as stage 4 cancer, frailty or severe COVID infections
25. Female who is pregnant or nursing
26. Current participation in another investigational drug or device treatment study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 48 hours post index procedure
  Change in RV/LV ratio
Safety: Composite of Major Adverse Device-Related Events | 48 hours post index procedure
  Device-related major bleeding at access, device-related death, clinical deterioration, pulmonary vascular injury or cardiac injury

SECONDARY OUTCOMES:
Safety: Composite of Major Adverse Events | 30 days post index procedure
  Assessment of major adverse events through 30 day follow-up

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (2):
  - Instituto do Coracao, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
- Dominican Republic (2):
  - Corazones Del Cibao, Santiago de los Caballeros, Santiago Province
  - Centro de Intervenciones Cardiovasculares, Santiago de los Caballeros, Santiago Province

IPD SHARING:
Plan to Share IPD: No